CLINICAL TRIAL: NCT02180308
Title: Lymph Node Assessment Using Simultaneous 18F-FDG-PET and MRI
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-00434
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Head and Neck Cancer
Keywords: Head cancer; Neck cancer; MRI; PET
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PET/MRI: Patient receives PET/MRI
  Interventions: Device: PET/MRI

INTERVENTIONS:
Device: PET/MRI — Simultaneous PET/MRI (3T system)
  Other Names: Siemens Biograph mMR

SUMMARY:
The overarching goal of this study is to develop PET/MR techniques to accurately detect nodal metastases for surgical planning and assessment of treatment response.

DETAILED DESCRIPTION:
Patients (n = 30) with head and neck cancer who are scheduled for node dissection surgery are eligible. Enrolled subjects will undergo one research PET/MR scan at the Center for Biomedical Imaging (660 First Avenue) within one week prior to the planned surgery. During the dissection, the locations of removed lymph nodes will be noted in terms of conventional neck lymph node levels. PET/MR data will be used for development of a combined kinetic model analysis of PET and MRI data (Aim 1). The final PET/MR findings will be compared with pathological evaluation results in order to assess the accuracy of PET/MR for detection of nodal metastases (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

Patients with head and neck cancer who are scheduled for node dissection surgeries at NYU Langone Medical Center or Bellevue hospital are eligible.

Exclusion Criteria:

Normal MRI exclusion criteria will apply, including those on the following list. A standard MRI safety form will be used to identify potential conditions warranting exclusion.

* Electrical implants such as cardiac pacemakers or perfusion pumps
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial heart, valves with steel parts, metal fragments, shrapnel, bullets, tattoos near the eye, or steel implants
* Ferromagnetic objects such as jewelry or metal clips in clothing
* Claustrophobia
* History of seizures
* Diabetes In addition, patients with GFR < 15 ml/min/1.73m2 or who are on dialysis will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck cancer who are scheduled for node dissection surgeries at NYU Langone Medical Center or Bellevue hospital.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Accuracy of simultaneous FDG-PET/MRI for detection of nodal metastases | 2 years after beginning of study (July 2014 - June 2016)
  This study is to assess PET/MR techniques for detection of nodal metastases for surgical planning and assessment of treatment response. Our central hypothesis is glucose metabolic rate (GMR) measured using a simultaneous PET/MR scanner can more accurately detect nodal metastases than standardized uptake value (SUV) measures from PET alone. SUV depends on both tumor metabolic rate and tracer delivery, which makes the interpretation of SUV challenging. For instance, an inflammatory node can have high SUV due to increased vascularity and vascular permeability and cannot be easily differentiated from a metastatic node, based on SUV. However, we hypothesize that inflammatory nodes will have lower GMR than metastatic nodes that contain highly proliferating cancer cells, such that they can be differentiated from metastatic nodes more reliably. This study will also determine if simultaneously acquired MRI can reduce uncertainty in GMR measurement of PET.

CONTACTS AND LOCATIONS:
Overall Officials: Sungheon Kim, PhD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States